CLINICAL TRIAL: NCT00379249
Title: Effects of a Twelve Months ROSUVASTATIN Treatment Plus Additional Care (Drug Intake Adherence and Lifestyle Enhancing Initiatives ) Compared to ROSUVASTATIN Treatment Alone on Long-Term Disease-Related Costs in Patients With an Indication for Statin Treatment According to the Joint European Guidelines
Brief Title: Rosuvastatin ORBITAL Germany
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D3560L00001; ORBITAL
Record Dates: First submitted 2006-09-20; First posted 2006-09-21 (Estimated); Last update posted 2009-03-26 (Estimated); Status verified 2009-03

CONDITIONS: Hypercholesterolemia
Keywords: hypercholesterolemia; statin; compliance
MeSH Terms: conditions — Hypercholesterolemia; Patient Compliance | interventions — Rosuvastatin Calcium

INTERVENTIONS:
Drug: Rosuvastatin

SUMMARY:
The primary objective of the study is to compare the effect of rosuvastatin therapy plus compliance initiatives and rosuvastatin therapy alone for 12 months (52 weeks) on long-term cumulative direct and indirect disease-related costs during the 36 month.

ELIGIBILITY:
Inclusion Criteria:

* high cholesterol with an indication for cholesterol-lowering medication (statins)

Exclusion Criteria:

* contra-indications for statin therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8000
Dates: Start 2002-02; Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
Cumulative direct/indirect disease-related costs were compared applying a societal perspective
Costs include resource utilization for ambulatory, hospital, rehabilitative and nursing care, medication, physiotherapy, transportation, and productivity loss)

SECONDARY OUTCOMES:
Achievement of the 1998 European LDL-C goal of <115 mg/dL (3.0 mmol/L)
Changes in the lipid profile and compliance with therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Meyer - Sabellek, MD, Study Director — AstraZeneca Germany; Stefan Stefan Willich, MD, Principal Investigator — Charité Berlin, Germany

REFERENCES:
- [Derived] Muckelbauer R, Englert H, Rieckmann N, Chen CM, Wegscheider K, Voller H, Katus HA, Willich SN, Muller-Nordhorn J. Long-term effect of a low-intensity smoking intervention embedded in an adherence program for patients with hypercholesterolemia: Randomized controlled trial. Prev Med. 2015 Aug;77:155-61. doi: 10.1016/j.ypmed.2015.05.026. Epub 2015 Jun 4. PMID 26051201
- [Derived] Muller-Nordhorn J, Muckelbauer R, Englert H, Grittner U, Berger H, Sonntag F, Voller H, Prugger C, Wegscheider K, Katus HA, Willich SN. Longitudinal association between body mass index and health-related quality of life. PLoS One. 2014 Mar 26;9(3):e93071. doi: 10.1371/journal.pone.0093071. eCollection 2014. PMID 24671104